CLINICAL TRIAL: NCT03777787
Title: The Relationship Between Acute Administration of a Bitter Compound and Transient Lower Esophageal Sphincter Relaxations and Reflux Events in Healthy Subjects
Brief Title: Bitter Tastants and Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: S61251
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Gastro Esophageal Reflux
Keywords: Bitter; TLESRs; Gastric tone
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — denatonium; Water

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bitter (Experimental): A single intragastric administration of denatonium benzoate (1 µmol/kg)
  Interventions: Dietary Supplement: Denatonium Benzoate
- Placebo (Placebo Comparator): A single intragastric administration of placebo (water)
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Denatonium Benzoate — A single intragastric administration of denatonium benzoate (1 µmol/kg)
  Arms: Bitter
Dietary Supplement: Water — A single intragastric administration of water
  Arms: Placebo

SUMMARY:
Recently the relationship between intragastric pressure (IGP) and reflux events after a meal was investigated, both in gastro-esophageal reflux disease (GERD) patients and in healthy volunteers. Ingestion of a meal was accompanied by a drop in IGP. However, the magnitude of this drop varied and was inversely correlated with the number of transient lower esophageal sphincter relaxations (TLESRs) and the number of reflux events, both in patients and in healthy volunteers: a smaller meal-induced drop in IGP was associated with a higher rate of reflux events and vice versa. This finding suggests that a smaller meal-induced drop may act as a trigger for reflux. It has been demonstrated that bitter administration leads to a smaller meal-induced drop. Therefore, bitter can be a dietary trigger for TLESRs facilitating the occurrence of symptoms of GERD. To evaluate this hypothesis, the researchers will study the relationship between bitter and the occurrence of TLESRs and reflux events in healthy volunteers. Additionally, it has been demonstrated that administering bitter also influences the concentration of motilin. Therefore, the research team will also measure the concentration of motilin to investigate whether changes in motilin concentrations can influence the number of TLESRs, via a change in gastric tone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers
* Age between 18 and 65
* Written informed consent

Exclusion Criteria:

* A history of any upper GI symptoms or GI surgery;
* Psychological disorders;
* Concomitant use of other medication or treatments except for oral contraceptives;
* Use of medication altering esophageal or GI motility;
* Pregnant or nursing women.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Change in number of TLESRs | 1 week
  Changes in the number of transient lower esophageal sphincter relaxations (TLESRs) between the placebo and bitter condition.

SECONDARY OUTCOMES:
Change in reflux | 1 week
  The change in the number of reflux events between placebo and bitter condition.
Change in motility pattern | 1 week
  The change in the intragastric pressure between placebo and bitter condition.
Change in motilin concentration | 1 week
  The change in motilin concentration between placebo and bitter condition.
Change in symptoms | 1 week
  Change in the number of volunteers reporting gastrointestinal symptoms between placebo and bitter condition

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium